CLINICAL TRIAL: NCT00574587
Title: Phase I-II Trial of Vorinostat Plus Weekly Paclitaxel (+/- Trastuzumab) Followed by Doxorubicin-cyclophosphamide in Patients With Locally Advanced Breast Cancer
Brief Title: Trial for Locally Advanced Breast Cancer Using Vorinostat Plus Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Joseph Sparano, Professor, Oncology, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-10-374; NYCC1 (Other: Montefiore Medical Center); NCI-2013-01216 (Registry Identifier: CTRP)
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Vorinostat; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Vorinostat; Paclitaxel; Trastuzumab; Doxorubicin; Cyclophosphamide; Surgical Procedures, Operative; Mastectomy; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat Plus Paclitaxel (Experimental): Vorinostat (PO days 1-3) plus weekly paclitaxel x 12 weeks (and trastuzumab if HER2-positive), followed by doxorubicin-cyclophosphamide every 2 weeks x 4 cycles, followed by surgery
  Interventions: Drug: Vorinostat; Drug: Paclitaxel; Drug: Trastuzumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Procedure: Surgery

INTERVENTIONS:
Drug: Vorinostat — Vorinostat 200 or 300 mg PO BID on days 1-3 of each weekly paclitaxel dose
  Other Names: Zolinza
Drug: Paclitaxel — Paclitaxel 80 mg/m2 weekly for 12 weeks
  Other Names: Taxol
Drug: Trastuzumab — Trastuzumab (if HER2-positive) 4 mg/kg, then 2 mg/kg weekly for 12 weeks including loading dose
  Other Names: Perception
Drug: Doxorubicin — Doxorubicin 60 mg/m2 every 2 weeks for 8 weeks
  Other Names: Adriamycin
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m2 every 2 weeks for 8 weeks
  Other Names: Cytoxan
Procedure: Surgery — Surgical excision of tumor from breast
  Other Names: Mastectomy or lumpectomy

SUMMARY:
Vorinostat is a histone deacetylase (HDAC) inhibitor which is approved by the U.S. Food and Drug Administration for the treatment of a rare type of cancer involving the skin (cutaneous T cell lymphoma), but not for breast cancer. HDAC inhibitors work by unsilencing tumor suppressor genes and other genes in the cancer cells that are repressed; when the genes are turned back on by the drug, it leads to death of the cancer cells. HDAC inhibitors such as vorinostat have been shown to enhance the effects of chemotherapy and trastuzumab in experimental systems. The purpose of this trial is to determine the optimal dose of vorinostat to use in combination with standard chemotherapy alone (or in combination with plus trastuzumab for HER2-positive disease), and to determine whether vorinostat enhances the effectiveness of standard chemotherapy (+/- trastuzumab) in patients with locally advanced breast cancer.

DETAILED DESCRIPTION:
This is a phase I-II trial in which patients with stage IIB-IIIC breast cancer will receive:

1. Neoadjuvant weekly paclitaxel (80 mg/m2 IV weekly x 12 weeks) plus vorinostat (200 or 300 mg PO BID on days 1-3 each paclitaxel dose) and trastuzumab (4 mg/kg loading dose, 2 mg/kg IV weekly x 12 total doses if HER2 positive, followed by:
2. Doxorubicin (60 mg/m2) plus cyclophosphamide (600 mg/m2) every 2 weeks x 4 cycles (plus G-CSF), followed by:
3. Surgery (lumpectomy or mastectomy)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast associated with the following stages: IIB, IIIA, IIIB or IIIC.
* Tumor must be Her2/neu positive
* No prior chemotherapy, radiation or definitive therapeutic surgery

Exclusion Criteria:

* May not be receiving any other investigational agents
* Uncontrolled intercurrent illness

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sparano, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: April 2008 - September 2013
Pre-assignment Details: Patients with HER2 positive disease also received trastuzumab.
Groups:
- Stratum A (HER2-positive): Dose Level 1: Vorinostat (PO days 1-3) plus weekly paclitaxel x 12 weeks and trastuzumab x 12 weeks, followed by doxorubicin-cyclophosphamide every 2 weeks x 4 cycles, followed by surgery
  Vorinostat: Vorinostat 200 mg PO BID on days 1-3 of each weekly paclitaxel dose
  Paclitaxel: Paclitaxel 80 mg/m2 weekly for 12 weeks
  Trastuzumab: Trastuzumab (if HER2-positive) 4 mg/kg, then 2 mg/kg weekly for 12 weeks including loading dose
  Doxorubicin: Doxorubicin 60 mg/m2 every 2 weeks for 8 weeks
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 every 2 weeks for 8 weeks
  Surgery: Surgical excision of tumor from breast
- Stratum A (HER2-positive): Dose Level 2; Stratum B: Triple Negative; Stratum C: ER-Positive, HER2-negative: Vorinostat (PO days 1-3) plus weekly paclitaxel x 12 weeks and trastuzumab x 12 weeks, followed by doxorubicin-cyclophosphamide every 2 weeks x 4 cycles, followed by surgery
  Vorinostat: Vorinostat 300 mg PO BID on days 1-3 of each weekly paclitaxel dose
  Paclitaxel: Paclitaxel 80 mg/m2 weekly for 12 weeks
  Trastuzumab: Trastuzumab (if HER2-positive) 4 mg/kg, then 2 mg/kg weekly for 12 weeks including loading dose
  Doxorubicin: Doxorubicin 60 mg/m2 every 2 weeks for 8 weeks
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 every 2 weeks for 8 weeks
  Surgery: Surgical excision of tumor from breast
Period: Overall Study
Arm/Group | Stratum A (HER2-positive): Dose Level 1 | Stratum A (HER2-positive): Dose Level 2 | Stratum B: Triple Negative | Stratum C: ER-Positive, HER2-negative
Started | 3 | 23 | 16 | 13
Completed | 3 | 23 | 16 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stratum A (HER2-positive): Dose Level 1: Vorinostat (PO days 1-3) plus weekly paclitaxel x 12 weeks and trastuzumab, followed by doxorubicin-cyclophosphamide every 2 weeks x 4 cycles, followed by surgery
  Vorinostat: Vorinostat 200 mg PO BID on days 1-3 of each weekly paclitaxel dose
  Paclitaxel: Paclitaxel 80 mg/m2 weekly for 12 weeks
  Trastuzumab: Trastuzumab (if HER2-positive) 4 mg/kg, then 2 mg/kg weekly for 12 weeks including loading dose
  Doxorubicin: Doxorubicin 60 mg/m2 every 2 weeks for 8 weeks
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 every 2 weeks for 8 weeks
  Surgery: Surgical excision of tumor from breast
- Stratum A (HER2-positive): Dose Level 2; Stratum B: Triple Negative; Stratum C: ER-Positive, HER2-Negative: Vorinostat (PO days 1-3) plus weekly paclitaxel x 12 weeks and trastuzumab, followed by doxorubicin-cyclophosphamide every 2 weeks x 4 cycles, followed by surgery
  Vorinostat: Vorinostat 300 mg PO BID on days 1-3 of each weekly paclitaxel dose
  Paclitaxel: Paclitaxel 80 mg/m2 weekly for 12 weeks
  Trastuzumab: Trastuzumab (if HER2-positive) 4 mg/kg, then 2 mg/kg weekly for 12 weeks including loading dose
  Doxorubicin: Doxorubicin 60 mg/m2 every 2 weeks for 8 weeks
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 every 2 weeks for 8 weeks
  Surgery: Surgical excision of tumor from breast
- Total: Total of all reporting groups
Arm/Group | Stratum A (HER2-positive): Dose Level 1 | Stratum A (HER2-positive): Dose Level 2 | Stratum B: Triple Negative | Stratum C: ER-Positive, HER2-Negative | Total
Number analyzed (Participants) | 3 | 23 | 16 | 13 | 55
Age, Continuous [Median (Full Range); unit: years] | 54 [30 to 69] | 54 [30 to 69] | 48 [41 to 64] | 46 [30 to 73] | 52 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 23 | 16 | 13 | 55
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose of Vorinostat in Combination With Weekly Paclitaxel/Trastuzumab
Description: Dose limiting toxicity in cycle 1
Time Frame: 3 weeks
Population: The recommended Phase II Dose of vorinostat was determined in Stratum A and B participants only.
Measure: Number; unit: mg
Groups:
- Stratum A: VR-Paclitaxel-Trastuzumab: Stratum A: Vorinostat 200 (Dose Level 1) or 300 mg (Dose level 2) by mouth on days 1-3 plus weekly paclitaxel 80 mg x 12 weeks and trastuzumab 4 mg/kg, then 2 mg/kg x 12 weeks, followed by doxorubicin 60 mg/m2 -cyclophosphamide 600 mg/m2 every 2 weeks x 8 weeks, followed by surgery
- Stratum B: VR-Paclitaxel-Trastuzumab: Stratum B: 300 mg by mouth on days 1-3 plus weekly paclitaxel 80 mg x 12 weeks and trastuzumab 4 mg/kg, then 2 mg/kg x 12 weeks, followed by doxorubicin 60 mg/m2 -cyclophosphamide 600 mg/m2 every 2 weeks x 8 weeks, followed by surgery
Arm/Group | Stratum A: VR-Paclitaxel-Trastuzumab | Stratum B: VR-Paclitaxel-Trastuzumab
Number analyzed (Participants) | 6 | 6
mg | 300 | 300

2. Secondary Outcome: Pathological Complete Response (CR) Rate in Patients With Her2/Neu Positive Locally Advanced Breast Cancer.
Description: Pathological Complete Response (CR) defined as absence of invasive cancer at surgery
Time Frame: 6 months
Population: Stratum A (HER2-positive): Dose Level 1 and Stratum A (HER2-positive): Dose Level 2 are combined. Data was collected for outcome measures per stratum not per dose level. 2 pts in Stratum A were not evaluable (1 lost to f/u; 1 death); 1 pt was not evaluable in Stratum B (1 death) and 1 pt was not evaluable in C (1 declined surgery)
Measure: Count of Participants; unit: Participants
Groups:
- Stratum A (HER2-positive): Vorinostat (PO days 1-3) plus weekly paclitaxel x 12 weeks and trastuzumab x 12 weeks, followed by doxorubicin-cyclophosphamide every 2 weeks x 4 cycles, followed by surgery
  Vorinostat: Vorinostat 200-300 mg PO BID on days 1-3 of each weekly paclitaxel dose
  Paclitaxel: Paclitaxel 80 mg/m2 weekly for 12 weeks
  Trastuzumab: Trastuzumab (if HER2-positive) 4 mg/kg, then 2 mg/kg weekly for 12 weeks including loading dose
  Doxorubicin: Doxorubicin 60 mg/m2 every 2 weeks for 8 weeks
  Cyclophosphamide: Cyclophosphamide 600 mg/m2 every 2 weeks for 8 weeks
  Surgery: Surgical excision of tumor from breast
Arm/Group | Stratum A (HER2-positive) | Stratum B: Triple Negative | Stratum C: ER-Positive, HER2-negative
Number analyzed (Participants) | 24 | 15 | 12
Participants | 13 | 4 | 0
Statistical Analysis 1: Comparison: Stratum A (HER2-positive) vs Stratum B: Triple Negative vs Stratum C: ER-Positive, HER2-negative; Test type: Superiority or Other; p < 0.10, Simon's Mimimax 2-stage design; 95% Confidence interval = 54, 20% CI 2-sided [34 to 74]

ADVERSE EVENTS:
Arm/Group | Stratum A (HER2-positive): Dose Level 1 | Stratum A (HER2-positive): Dose Level 2 | Stratum B: Triple Negative | Stratum C: ER-Positive, HER2-negative
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/23 | 1/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/23 | 1/16 | 0/13
Other Adverse Events (participants affected / at risk) | 0/3 | 0/23 | 0/16 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (HER2-positive): Dose Level 1 (N=3) | Stratum A (HER2-positive): Dose Level 2 (N=23) | Stratum B: Triple Negative (N=16) | Stratum C: ER-Positive, HER2-negative (N=13)
pulmonary emobolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No